CLINICAL TRIAL: NCT00801671
Title: Study of Independent Role of Continuous Positive Airway Pressure Therapy on Systemic Arterial Pressure in Patients With Sleep Apnea Syndrome and Arterial Hypertension
Brief Title: Russian Study of the Effect of Continuous Positive Airway Pressure (CPAP) in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Russian Cardiology Research and Production Center (Other)
Responsible Party: Kseniya Orlowa, Weinmann
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2008-06-19; First posted 2008-12-03 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Obstructive Sleep Apnea Syndrome; Hypertension
Keywords: obstructive sleep apnea; obstructive sleep apnea syndrome; hypertension; systemic hypertension; ambulatory blood pressure monitoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: cPAP
- 2 (Sham Comparator)
  Interventions: Procedure: cPAP

INTERVENTIONS:
Procedure: cPAP — After reaching target level of BP patients will be randomized in active group (cPAP) and control group (sham-cPAP)

SUMMARY:
The purpose of this study is to determine whether CPAP is effective in the treatment of systemic hypertension.

DETAILED DESCRIPTION:
It is now well known that cardiovascular risks are increased in patients with obstructive sleep apnea syndrome (OSAS). Also a link has already been demonstrated between OSAS and hypertension.

Nowadays, the most efficient treatment of the OSAS is the continuous Positive Airway Pressure (cPAP). Several studies have also shown that cPAP could reduce arterial blood pressure in OSAS patients. But level of blood pressure (BP), drug treatment were not equal between groups and it's difficult to single out independent role of cPAP.

Our study has the objective to compare the effects of cPAP on hypertension in OSAS patients. After 3-9 weeks of antihypertensive treatment (valsartan and amlodipine) those one who reached target level of BP will be randomized either in the group "treatment by cPAP" or in the group "treatment by cham-cPAP" for 3 weeks and then we'll perform cross-over.

ELIGIBILITY:
Inclusion Criteria:

* male/female over than 18 years old
* patient with an obstructive sleep apnea (apnea-hypopnea index > or equal to 15)
* patient with weak or moderate hypertension (140 <= SBP < 180 mmHg and 90 <= DBP < 110 mmHg)
* negative pregnancy test
* ambulatory patient
* patient who have signed the informed consent form

Exclusion Criteria:

* pregnant or nursing woman
* woman who refuses to use contraceptive method
* acute hepatic failure, biliary cirrhosis, cholestasis
* clearance of Cockcroft < 30 ml/min/1.73m2
* kaliemia >= 5.5 mmol/l
* acute hypertension (SBP>= 180 mmHg and/or DBP >= 110 mmHg)
* acute daytime sleepiness (Epworth rating scale > 15)
* patient with a profession that is inconsistent with the continuous positive airway pressure (CPAP) treatment
* known cardiovascular pathologies
* contraindication to CPAP
* allergy to valsartan and/or amlodipine
* patient treated with lithium
* patient on tutelle or curatelle
* patient kept in detention, major protected by the law, hospitalized person patient currently participating in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure monitoring over 24 hours, at inclusion visit (day=0), before cPAP (3-9 weeks) and after 3 weeks of cPAP. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexandr Yu Litvin, MD, Principal Investigator — Russian Cardiology Research and Production Center
Locations (1):
- Russian Cardiologe Research and Production Complex, Moscow, Russia

REFERENCES:
- [Derived] Litvin AY, Sukmarova ZN, Elfimova EM, Aksenova AV, Galitsin PV, Rogoza AN, Chazova IE. Effects of CPAP on "vascular" risk factors in patients with obstructive sleep apnea and arterial hypertension. Vasc Health Risk Manag. 2013;9:229-35. doi: 10.2147/VHRM.S40231. Epub 2013 May 10. PMID 23690688